CLINICAL TRIAL: NCT01964222
Title: A Mixed Methods Study to Reduce Disparities in Cancer Clinical Trials by Adapting a Health Literacy Intervention for Informed Consent and Comparing it to Usual Care in a Randomized Experiment
Brief Title: Health Literacy Intervention for Informed Consent of Cancer Patients Considering Clinical Trial Participation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 201309076
Record Dates: First submitted 2013-10-07; First posted 2013-10-17 (Estimated); Results first posted 2015-12-07 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-11

CONDITIONS: Cancer
Keywords: Cancer; Clinical trials; Informed consent; Health literacy
MeSH Terms: conditions — Neoplasms | interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Decision Aid (DA) (Experimental): The decision aid (DA) will be provided to patients randomized to the experimental/intervention group.
  Interventions: Behavioral: Decision Aid (DA)
- Control (No Intervention): Participants randomized to the control group will receive usual care and will be shown Siteman Cancer Center website about clinical trials.

INTERVENTIONS:
Behavioral: Decision Aid (DA) — Participants will be shown (on a computer) a targeted, web-based decision aid focused on the topic of clinical trials in addition to usual care.
  Arms: Decision Aid (DA)

SUMMARY:
This study will update an existing health literacy intervention (decision aid) for informed consent procedures and then conduct a randomized experiment implementing the health literacy intervention at Siteman Cancer Center and evaluate its effectiveness compared to usual care. Our hypothesis is that implementing the targeted, web-based decision aid (DA) in addition to usual care will increase knowledge about cancer clinical trials. Secondary outcomes include patients' ability to communicate with health care providers about trials, willingness to participate in trials, and enrollment rates for minority participants.

DETAILED DESCRIPTION:
A previously developed and pilot tested web-based decision aid (DA) based on best practices in health literacy that is well received by minority participants and significantly improved knowledge about cancer clinical trials and decision self-efficacy will be used. This study will expand the reach of the DA and test it in a larger study in a different geographic region and center (Siteman Cancer Center). An additional benefit of conducting this work at Siteman Cancer Center is that Siteman and the Program for the Elimination of Cancer Disparities (PECaD) already institute structural changes at the system level to improve minority participation in trials. This study will activate and educate patients and will complement the system-level interventions.

By random 1:1 assignment, 180 participants will either receive:

*Targeted, web-based decision aid (DA) about participating in cancer clinical trials.

or

*Usual care/control-Access to the Siteman Cancer Center website about clinical trials.

Outcomes from the DA group will be compared to outcomes in a usual care/control group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cancer in the past 6 months
* English speaking
* At least 18 years old

Exclusion Criteria:

* Past participation in a clinical trial for treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2014-05; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary C Politi, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Siteman Cancer Center, St Louis, Missouri, United States

REFERENCES:
- [Background] Murthy VH, Krumholz HM, Gross CP. Participation in cancer clinical trials: race-, sex-, and age-based disparities. JAMA. 2004 Jun 9;291(22):2720-6. doi: 10.1001/jama.291.22.2720. PMID 15187053
- [Background] Janet Yang Z, McComas K, Gay G, Leonard JP, Dannenberg AJ, Dillon H. From information processing to behavioral intentions: exploring cancer patients' motivations for clinical trial enrollment. Patient Educ Couns. 2010 May;79(2):231-8. doi: 10.1016/j.pec.2009.08.010. Epub 2009 Sep 11. PMID 19748204
- [Background] Institute of Medicine (US) Committee on Assessing the System for Protecting Human Research Participants; Federman DD, Hanna KE, Rodriguez LL, editors. Responsible Research: A Systems Approach to Protecting Research Participants. Washington (DC): National Academies Press (US); 2002. Available from http://www.ncbi.nlm.nih.gov/books/NBK43563/ PMID 20669487
- [Background] Silverman H, Hull SC, Sugarman J. Variability among institutional review boards' decisions within the context of a multicenter trial. Crit Care Med. 2001 Feb;29(2):235-41. doi: 10.1097/00003246-200102000-00002. PMID 11246299
- [Background] McNutt LA, Waltermaurer E, Bednarczyk RA, Carlson BE, Kotval J, McCauley J, Campbell JC, Ford DE. Are We Misjudging How Well Informed Consent Forms are Read? J Empir Res Hum Res Ethics. 2008 Mar;3(1):89-97. doi: 10.1525/jer.2008.3.1.89. PMID 19385786
- [Background] Grossman SA, Piantadosi S, Covahey C. Are informed consent forms that describe clinical oncology research protocols readable by most patients and their families? J Clin Oncol. 1994 Oct;12(10):2211-5. doi: 10.1200/JCO.1994.12.10.2211. PMID 7931491
- [Background] Corbie-Smith G, Thomas SB, Williams MV, Moody-Ayers S. Attitudes and beliefs of African Americans toward participation in medical research. J Gen Intern Med. 1999 Sep;14(9):537-46. doi: 10.1046/j.1525-1497.1999.07048.x. PMID 10491242
- [Background] Featherstone K, Donovan JL. Random allocation or allocation at random? Patients' perspectives of participation in a randomised controlled trial. BMJ. 1998 Oct 31;317(7167):1177-80. doi: 10.1136/bmj.317.7167.1177. PMID 9794849
- [Background] Joffe S, Cook EF, Cleary PD, Clark JW, Weeks JC. Quality of informed consent in cancer clinical trials: a cross-sectional survey. Lancet. 2001 Nov 24;358(9295):1772-7. doi: 10.1016/S0140-6736(01)06805-2. PMID 11734235
- [Background] Dresden GM, Levitt MA. Modifying a standard industry clinical trial consent form improves patient information retention as part of the informed consent process. Acad Emerg Med. 2001 Mar;8(3):246-52. doi: 10.1111/j.1553-2712.2001.tb01300.x. PMID 11229946
- [Background] Young DR, Hooker DT, Freeberg FE. Informed consent documents: increasing comprehension by reducing reading level. IRB. 1990 May-Jun;12(3):1-5. No abstract available. PMID 11651387
- [Background] Krumholz HM. Informed consent to promote patient-centered care. JAMA. 2010 Mar 24;303(12):1190-1. doi: 10.1001/jama.2010.309. No abstract available. PMID 20332406
- [Background] Coyne CA, Xu R, Raich P, Plomer K, Dignan M, Wenzel LB, Fairclough D, Habermann T, Schnell L, Quella S, Cella D; Eastern Cooperative Oncology Group. Randomized, controlled trial of an easy-to-read informed consent statement for clinical trial participation: a study of the Eastern Cooperative Oncology Group. J Clin Oncol. 2003 Mar 1;21(5):836-42. doi: 10.1200/JCO.2003.07.022. PMID 12610182
- [Background] Davis TC, Holcombe RF, Berkel HJ, Pramanik S, Divers SG. Informed consent for clinical trials: a comparative study of standard versus simplified forms. J Natl Cancer Inst. 1998 May 6;90(9):668-74. doi: 10.1093/jnci/90.9.668. PMID 9586663
- [Background] Flory J, Emanuel E. Interventions to improve research participants' understanding in informed consent for research: a systematic review. JAMA. 2004 Oct 6;292(13):1593-601. doi: 10.1001/jama.292.13.1593. PMID 15467062
- [Background] Entwistle V. Supporting participation in clinical research: decision aids for trial recruitment? Health Expect. 2008 Sep;11(3):205-7. doi: 10.1111/j.1369-7625.2008.00519.x. No abstract available. PMID 18816317
- [Background] Brehaut JC, Lott A, Fergusson DA, Shojania KG, Kimmelman J, Saginur R. Can patient decision aids help people make good decisions about participating in clinical trials? A study protocol. Implement Sci. 2008 Jul 23;3:38. doi: 10.1186/1748-5908-3-38. PMID 18651981
- [Background] Byrne MM, Tannenbaum SL, Gluck S, Hurley J, Antoni M. Participation in cancer clinical trials: why are patients not participating? Med Decis Making. 2014 Jan;34(1):116-26. doi: 10.1177/0272989X13497264. Epub 2013 Jul 29. PMID 23897588
- [Background] Sutherland HJ, da Cunha R, Lockwood GA, Till JE. What attitudes and beliefs underlie patients' decisions about participating in chemotherapy trials? Med Decis Making. 1998 Jan-Mar;18(1):61-9. doi: 10.1177/0272989X9801800113. PMID 9456210
- [Background] Office of Human Research Protections (OHRP): Compliance Determination Letters. US Department of Health and Human Services. Washington, DC: 2002.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Decision Aid (DA) | Control
Started | 101 | 100
Completed | 86 | 89
Not Completed | 15 | 11
Not completed — Lost to Follow-up | 7 | 5
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Screening Failure | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Decision Aid (DA) | Control | Total
Number analyzed (Participants) | 86 | 89 | 175
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.81 (12.26) | 53.88 (12.05) | 54.83 (12.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 68 | 132
  Male | 22 | 21 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 85 | 86 | 171
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 5
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 18 | 35
  White | 64 | 66 | 130
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Rapid Estimate of Adult Literacy in Medicine-SF (REALM-SF) [Number; unit: participants] — 5 participants did not complete this measure due to lack of time during enrollment.
  participants
    Inadequate | 5 | 5 | 10
    Marginal | 20 | 13 | 33
    Adequate | 61 | 66 | 127

OUTCOME MEASURES:

1. Primary Outcome: Knowledge About Cancer Clinical Trials
Description: A questionnaire will be administered to assess outcomes of interest immediately after showing the participant either the decision aid (DA) about clinical trials or the Siteman Cancer Center website about clinical trials. The questionnaire will include eleven knowledge items such as "Only very sick patients are asked to take part in a cancer research study" and "Cancer research studies almost never involve the use of a placebo or sugar pill alone". Participants will indicate each item as "True", "False", or "I don't know". An overall knowledge composite score will be created with the average percentage of items participants in each condition correctly answer. Participation in study concludes upon completion of questionnaire.
Time Frame: 1 day (Immediately following either showing the participant the experimental or control information (same day)
Population: Analysis is represented as mean (standard deviation) of percentage of knowledge questions answered correctly.
Measure: Mean (Standard Deviation); unit: percentage questions answered correctly
Arm/Group | Decision Aid (DA) | Control
Number analyzed (Participants) | 86 | 89
percentage questions answered correctly | 73.4 (21.6) | 61.6 (18.8)

2. Secondary Outcome: Self-efficacy for Communicating About Cancer Clinical Trials
Description: A questionnaire will be administered to assess outcomes of interest immediately after showing the participant either the decision aid (DA) about clinical trials or the Siteman Cancer Center website about clinical trials. The questionnaire will include an item in which participants rank their self-efficacy for finding information about cancer clinical trials on a 5-point scale with higher numbers indicating greater self-efficacy. Participation in study concludes upon completion of questionnaire.
Time Frame: 1 day (Immediately following either showing the participant the experimental or control information (same day)
Population: Analysis is represented as mean (standard deviation) of participant-reported self-efficacy for finding information about cancer clinical trials.
Measure: Mean (Standard Deviation); unit: units on a scale of 1 to 5
Arm/Group | Decision Aid (DA) | Control
Number analyzed (Participants) | 86 | 89
units on a scale of 1 to 5 | 4.1 (1.0) | 3.5 (1.1)

3. Primary Outcome: Clarity of Values
Description: A questionnaire will be administered to assess outcomes of interest immediately after showing the participant either the decision aid (DA) about clinical trials or the Siteman Cancer Center website about clinical trials. The questionnaire will include the Values Clarity Subscale to evaluate decisional conflict. The subscale includes two items from the ten-item Low Literacy Decisional Conflict Scale, each with three response categories. The combined score on the two items will be divided by 2 and multiplied by 25 to produce an overall "values clarity" score from 0 to 100. Higher values represent less clarity. Participation in study concludes upon completion of questionnaire.
Time Frame: 1 day (Immediately following either showing the participant the experimental or control information (same day)
Population: Analysis is represented as mean (standard deviation) of calculated values clarity.
Measure: Mean (Standard Deviation); unit: units on a scale of 0 to 100
Arm/Group | Decision Aid (DA) | Control
Number analyzed (Participants) | 86 | 89
units on a scale of 0 to 100 | 16.6 (27) | 33 (36.5)

4. Primary Outcome: Uncertainty in Choice
Description: A questionnaire will be administered to assess outcomes of interest immediately after showing the participant either the decision aid (DA) about clinical trials or the Siteman Cancer Center website about clinical trials. The questionnaire will include the Uncertainty Subscale to evaluate decisional conflict. The subscale includes two items from the ten-item Low Literacy Decisional Conflict Scale, each with three response categories. The combined score on the two items will be divided by 2 and multiplied by 25 to produce an overall "uncertainty" score from 0 to 100. Higher values represent more uncertainty. Participation in study concludes upon completion of questionnaire.
Time Frame: 1 day Immediately following either showing the participant the experimental or control information (same day)
Population: Analysis is represented as mean (standard deviation) of calculated uncertainty.
Measure: Mean (Standard Deviation); unit: units on a scale of 0 to 100
Arm/Group | Decision Aid (DA) | Control
Number analyzed (Participants) | 86 | 89
units on a scale of 0 to 100 | 23 (30.3) | 33.2 (33.2)

5. Secondary Outcome: Attitudes About Cancer Clinical Trials
Description: A questionnaire will be administered to assess outcomes of interest immediately after showing the participant either the decision aid (DA) about clinical trials or the Siteman Cancer Center website about clinical trials. The questionnaire will include two items in which participants rank their intent to participate in a cancer clinical trial and their intent to encourage others to participate in a cancer clinical trial on a 5-point scale with higher numbers indicating greater intent. Participation in study concludes upon completion of questionnaire.
Time Frame: 1 day (Immediately following either showing the participant the experimental or control information (same day)
Population: Analysis is represented as mean (standard deviation) of participant-reported intent.
Measure: Mean (Standard Deviation); unit: units on a scale of 1 to 5
Arm/Group | Decision Aid (DA) | Control
Number analyzed (Participants) | 86 | 89
units on a scale of 1 to 5
  Intent to Participate | 3.8 (1.1) | 3.8 (1.1)
  Intent to Encourage Others to Particpate | 3.7 (1.1) | 3.7 (1.0)

ADVERSE EVENTS:
Description: "Serious" and "Other" adverse events were not collected/assessed.
Arm/Group | Decision Aid (DA) | Control
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No